CLINICAL TRIAL: NCT01549366
Title: A Multi-Center Prospective Randomized Study Comparing Supplemental Posterior Instrumentation, Aspen™ Spinous Process System Versus Pedicle Screw Fixation, in Lateral Lumbar Interbody Fusion (LLIF) or Anterior Lumbar Interbody Fusion (ALIF)
Brief Title: Comparison of the Aspen Device Versus Pedicle Screws for Supplemental Posterior Fixation in Lumbar Interbody Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-11-001
Record Dates: First submitted 2012-02-29; First posted 2012-03-09 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
MeSH Terms: interventions — Pedicle Screws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspen Spinous Process Fixation Device (Experimental): Subjects randomized to the Aspen study arm will have the Aspen device implanted as supplemental posterior fixation only and according to the manufacturer's recommendations.
  Interventions: Device: Aspen Spinous Process Fixation Device
- Pedicle Screws (Active Comparator): Subjects randomized to the pedicle screw group will have polyaxial top loading pedicle screws implanted according to the standard procedures and practices at that institution. The procedure may be performed according to surgeon preference, including a traditional open, minimally invasive or percutaneous approach. Only pedicle screws cleared by FDA for this indication will be used in this study.
  Interventions: Device: Pedicle Screws

INTERVENTIONS:
Device: Aspen Spinous Process Fixation Device — The Aspen device will be placed as posterior fixation to Lateral Lumbar Interbody Fusion (LLIF) or Anterior Lumbar Interbody Fusion (ALIF)
  Arms: Aspen Spinous Process Fixation Device
Device: Pedicle Screws — Pedicle Screws will be placed as posterior fixation to Lateral Lumbar Interbody Fusion (LLIF) or Anterior Lumbar Interbody Fusion (ALIF)
  Arms: Pedicle Screws

SUMMARY:
The purpose of this clinical investigation is to evaluate the Aspen™ device compared to pedicle screw instrumentation for posterior fixation in the treatment of patients with degenerative disc disease and/or spondylolisthesis. The Aspen™ device will be compared to pedicle screw instrumentation in Oswestry Disability Index (ODI) improvement and success of fusion.

DETAILED DESCRIPTION:
This is a multi-center, prospective randomized clinical study to evaluate the clinical outcome of subjects with degenerative disc disease (DDD) (defined as back pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies) and/or spondylolisthesis utilizing either Aspen Spinous Process Fixation System or Pedicle Screws for supplemental posterior instrumentation as an adjunct to an anterior or lateral approach to lumbar interbody fusion.

The primary hypothesis is that change in Oswestry Disability Index (ODI) of subjects in the study group (Aspen) will be non-inferior to the control group (pedicle screw instrumentation). The non-inferiority margin is pre-specified to be 10 ODI score points. If the non-inferiority is established, superiority of Aspen to the control will be tested.

The study will involve up to 25 investigational sites. Enrollment is expected to take approximately 24 months. Subjects will be followed for 2 years, with the anticipated duration of the study being approximately 4 years from start to finish.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Scheduled for an elective single-level circumferential lumbar fusion by means of supplemental posterior fusion with fixation (allowing for the placement of ASPEN or pedicle screws) for an anterior or lateral interbody fusion
* Diagnosis of primary symptomatic Degenerative Disc Disease (DDD) and/or spondylolisthesis confirmed with appropriate imaging studies and/or positive lumbar discography
* Oswestry Disability Index (ODI) v2.1 score > 30%
* Failed at least 3 months of conservative care (non-surgical) OR has clinical signs of neurological deterioration
* Signed Informed Consent Form

Exclusion Criteria:

* Previous fusion at the operative level
* Spondylolisthesis Grade 3 or more
* Lytic spondylolisthesis
* Incompetent or missing posterior arch at the affected level (e.g. complete laminectomy, pars defect)
* Requires complete laminectomy at level of surgery
* Facet joints at implant level are absent or fractured
* Vertebral body compromise or acute fracture at implant level
* Body mass Index (BMI) ≥ 35
* Known allergy to titanium
* Osteoporosis: Simple Calculated Osteoporosis Risk Estimation (S.C.O.R.E.) > 6 AND Dual-energy X-ray absorptiometry (DEXA) T-score < -2.5
* Paget's disease, osteomalacia, or any other metabolic bone disease
* Use of medications or any drug known to potentially interfere with bone/soft tissue healing (e.g. chronic systemic steroids)
* Planned use of additional segmental fixation (eg. facet screws)
* Planned use of Bone Morphogenetic Protein (BMP) for posterolateral fusion*
* Unlikely to comply with the follow-up evaluation schedule
* In the opinion of the Investigator, Subject has history of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation
* Active participation in a clinical trial of another drug or device
* Active systemic infection or any other health condition that would preclude surgery
* History of invasive malignancy, except if the subject has received treatment and displayed no clinical signs and symptoms for at least five years
* Subject is a prisoner
* Pregnant or planning to become pregnant during the length of study participation
* Involvement in active litigation related to back problems at the time of screening
* Direct involvement in the execution of this protocol
* Pre-existing conditions that could interfere with the evaluation of outcome measures (e.g. musculoskeletal, neuromuscular, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Absolute change in Oswestry Disability Index (ODI) | baseline to 12 months post-operative

SECONDARY OUTCOMES:
Fusion success | 12 months and 24 months
Neurological status | Baseline, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Change in EQ-5D-3L | Baseline, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Change in SF-36 | Baseline, 12 months & 24 months
Change in Visual Analogue Scale (VAS) (pain) | Baseline, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Change in Zurich Claudication Questionnaire | Baseline, 12 months & 24 months
Pain medication usage | Baseline, surgery, 6 weeks, 3 months, 6 months, 12 months, & 24 months
Operative parameters (estimate blood loss, fluor time, length of hospital stay) | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Patel, Principal Investigator — University of Colorado, Denver; Cappuccino, Principal Investigator — Buffalo Spine Surgery
Locations (3):
- United States (3):
  - Clint Hill, Paducah, Kentucky
  - Buffalo Spine Surgery, Lockport, New York
  - Andy Kranenburg, Medford, Oregon

IPD SHARING:
Plan to Share IPD: Undecided